CLINICAL TRIAL: NCT00406731
Title: Role of endothelin-and Nitric Oxide-system in the Regulation of Optic Nerve Head Blood Flow During Changes in Ocular Perfusion Pressure
Brief Title: Role of Endothelin- and Nitric Oxide-system in the Regulation of Optic Nerve Head Blood Flow During Changes in Ocular Perfusion Pressure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OPHT-080206
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Ocular Physiology; Optic Disk; Regional Blood Flow
Keywords: Endothelin-1; L-NG-Monomethyl Arginine; Optic Nerve Head blood flow
MeSH Terms: interventions — omega-N-Methylarginine; Endothelin-1; Laser-Doppler Flowmetry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: NG-monomethyl-L-arginine (L-NMMA) — bolus 6 mg/kg over 5 minutes followed by a continuous intravenous infusion of 60 µg/kg/min over 12 minutes; twice on 1 study day
Drug: Endothelin-1 (ET-1) — 5 ng/kg/min intravenous infusion over 17 minutes; twice on 1 study day
Drug: Physiologic saline solution (placebo control) — intravenous infusion over 20 minutes; twice on 1 study day
Device: Laser Doppler flowmetry — blood flow measurements at the temporal neuroretinal rim of the optic nerve head
Device: Goldmann applanation tonometer — Intraocular pressure measurements
Device: HP-CMS patient monitor — blood pressure and pulse rate measurements
Procedure: Suction cup method — The IOP will be raised by an 11 mm diameter, standardized suction cup placed on the temporal sclera with the anterior edge at least 1 mm from the limbus.

SUMMARY:
Autoregulation is the ability of a vascular bed to maintain blood flow despite changes in perfusion pressure. The existence of an effective autoregulation in the optic nerve circulation has been shown in animals and humans. The exact mechanism behind this autoregulation is still unknown. The motive for the investigation of optic nerve head (ONH) blood flow autoregulation is to enhance the understanding of pathologic eye conditions associated with ocular vascular disorders. To clarify the regulatory mechanisms of ONH microcirculation is of critical importance to understand the pathophysiology of glaucoma because there is evidence that glaucoma is associated with optic nerve head ischemia. Several studies indicate that a disturbed autoregulation might contribute to glaucomatous optic neuropathy. Previous findings suggest endothelial dysfunction in glaucomatous optic neuropathy, in particular alterations in endothelin- and nitric oxide- system, which both play an important role in local regulation of vascular tone.

In the present study, changes in ocular perfusion pressure will be performed during administration of drugs, which may potentially alter the pressure-flow relationship. These drugs include endothelin-1 and the nitric oxide synthase inhibitor NG-monomethyl-L-arginine (L-NMMA).

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile (Must et al. 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 1 Dpt

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of systemic or pulmonary hypertension, or other cardiac or pulmonary diseases
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
ONH pressure-flow relationship | up to 3 study days

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, MD,Univ.Doz., Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria